CLINICAL TRIAL: NCT06329258
Title: A Single Center Study to Evaluate the Effectiveness and Safety of SOTYKTU® (Deucravacitinib) in Combination With Enstilar® for Moderate to Severe Plaque Psoriasis
Brief Title: Combination of Sotyktu and Enstilar for Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC09
Record Dates: First submitted 2024-03-14; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — betamethasone dipropionate, calcipotriol drug combination; calcipotriene; Betamethasone; deucravacitinib

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deucravacitinib in combination with Enstilar (Experimental): deucravacitinib in combination with Enstilar
  Interventions: Drug: Enstilar; Drug: Deucravacitinib
- Deucravacitinib monotherapy (Experimental): monotherapy
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Enstilar — Add on Enstilar
  Other Names: calcipotriene and betamethasone
  Arms: Deucravacitinib in combination with Enstilar
Drug: Deucravacitinib — 6mg QD
  Other Names: Sotyktu

SUMMARY:
combination deucravacitinib and enstilar foam

DETAILED DESCRIPTION:
30 adult patients with moderate to severe plaque psoriasis will be given Deucravacitinib 6mg QD for the first 8 weeks of the study.

At week 8:

Subjects who do not meet PASI 25 at week 8 will be discontinued from the study as non-responders.

Subjects who achieve ≥PASI 75 at week 8 will remain enrolled and continue Deucravacitinib 6mg QD monotherapy through week 24.

Subjects who achieved between PASI 25-74 response will receive 4 weeks of Enstilar (calcipotriene and betamethasone dipropionate) Foam, 0.005%/0.064% applied QD in addition to continuing Deucravacitinib 6mg QD.

At week 12, (after 4 consecutive weeks of Enstilar), subjects in the PASI 25-74 group, will discontinue Enstilar QD and continue Deucravacitinib as monotherapy through week 24.

Subjects will return at week 28 for safety follow evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult ≥ 18 years of age;
2. Diagnosis of chronic plaque-type psoriasis
3. Moderate to severe plaque type psoriasis as defined at baseline by:

   * BSA affected by plaque-type psoriasis of 10% or greater
   * PGA score of 3 or greater
   * PASI ≥ 12.
4. Able and willing to give written informed consent prior to performance of any study-related procedures Must be in general good health (except for disease under study) as judged by the Investigator, based on medical history, physical examination, clinical laboratories, and urinalysis.

Exclusion Criteria:

1. Other than psoriasis, any clinically significant (as determined by the investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is uncontrolled.
2. Forms of psoriasis other than chronic plaque-type (e.g., Pustular erythrodermic and/or guttate psoriasis) or drug induced psoriasis
3. Use of oral systemic medications or PUVA phototherapy for the treatment of psoriasis within 4 weeks (includes, but not limited to, oral corticosteroids, methotrexate, acitretin and cyclosporine).
4. Prior use of biologics within the following periods:

   * Etanercept - 4 weeks
   * Adalimumab or certolizumab pegol - 8 weeks
   * IL-17 antagonists - 16 weeks
   * Ustekinumab or IL-23 pathway inhibitors - 24 weeks
   * Other biologics - 5 half-lives
5. Patient used topical therapies or UVB phototherapy to treat psoriasis within 2 weeks of the Baseline Visit (includes, but not limited to, topical corticosteroids, vitamin D analogs, or retinoids).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index 75 at week 12 | 12 weeks
  Proportion of subjects achieving PASI 75 at week 12 for patients in the Deucravacitinib + Enstilar combination arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Schweiger Derm Group, East Windsor, New Jersey, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT06329258/Prot_SAP_000.pdf